CLINICAL TRIAL: NCT03998670
Title: Intermittent Exotropia Study 6: A Pilot Randomized Clinical Trial of Base-in Prism Spectacles for Intermittent Exotropia
Brief Title: Base-in Prism Spectacles for Intermittent Exotropia
Acronym: IXT6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Pediatric Eye Disease Investigator Group (Network); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IXT6; 2UG1EY011751 (NIH)
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Results first posted 2022-10-17 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Exotropia Intermittent
Keywords: Prism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: At the 8-week outcome visit, a Masked Examiner, who is a pediatric ophthalmologist, pediatric optometrist, or certified orthoptist, will assess the control of the exodeviation and perform PACT testing. The Masked Examiner must be someone other than the investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prism Group (Experimental): Spectacles with refractive correction and base-in relieving prism (40% of the greater of the exodeviation by prism and alternate cover test (PACT) at distance or near) equally divided between the 2 lenses will be prescribed to the participant
  Interventions: Device: Prism Glasses
- Non-Prism Group (Placebo Comparator): Spectacles with refractive correction (or plano spectacles if no significant refractive error) and no prism will be prescribed to the participant
  Interventions: Device: Non-Prism Glasses

INTERVENTIONS:
Device: Prism Glasses — Spectacles with refractive correction and base-in relieving prism (40% of the greater of the exodeviation by PACT at distance or near) equally divided between the 2 lenses
  Arms: Prism Group
Device: Non-Prism Glasses — Spectacles with refractive correction (or plano spectacles if no significant refractive error) and no prism
  Arms: Non-Prism Group

SUMMARY:
The objective of this short-term, pilot randomized trial comparing spectacles with relieving prism to spectacles without prism is to determine whether to proceed to a full-scale, longer-term randomized trial. This decision will be based primarily on assessing the initial (8-week) response to prism by comparing treatment groups on the following outcomes:

* Mean distance intermittent exotropia (IXT) control score (the mean of 3 control scores) (primary outcome)
* The proportion of participants demonstrating a "treatment response," defined as ≥1 point improvement in the mean distance IXT control score without spontaneous exotropia during control testing (secondary outcome)
* The proportion of participants reporting adverse effects and good/excellent spectacle wear compliance

ELIGIBILITY:
Inclusion Criteria:

Intermittent Exotropia meeting all of the following criteria:

* Age 3 to 13 years
* Mean distance control score of ≥2.00 points with at least 1 measure of 3, 4, or 5 points (i.e, spontaneous tropia) from the 3 assessments during the exam
* A near control score ≤4 on at least 1 of 3 assessments (cannot have score of 5, 5, 5)
* Distance exodeviation between 16 Prism Diopters (Δ) and 35 Δ (inclusive) by PACT
* Near exodeviation between 10 Δ and 35 Δ (inclusive) by PACT
* Near deviation does not exceed distance deviation by more than 10 Δ by PACT (i.e., convergence insufficiency-type IXT excluded)
* Refractive error between -6.00 Diopters (D) spherical equivalent (SE) and +2.50 D SE (inclusive) (based on a cycloplegic refraction performed within 7 months but prior to the day of enrollment)
* Refractive correction (must be worn for at least 1 week if refractive error meets any of the following (based on a cycloplegic refraction performed within 7 months but prior to the day of enrollment):

  * SE anisometropia ≥1.00 D
  * Astigmatism ≥1.00 D in either eye
  * SE myopia ≥-0.50 D in either eye
* If spectacles have been prescribed and are worn, they must meet the following pre- enrollment criteria:

  * SE anisometropia corrected to within 1.00 D of full SE anisometropic difference
  * Astigmatism corrected to within 1.00 D of full magnitude; axis within 10 degrees if astigmatism ≤1.00 D and axis within 5 degrees if astigmatism >1.00 D

Exclusion Criteria:

* Dissociated vertical deviation (DVD)
* Vertical deviation >3 Δ in primary gaze at distance or near
* Patterns (such as an "A" or "V" pattern) with a downgaze measurement of >10 Δ difference from straight ahead by PACT, measured per investigator's routine method
* Treatment for IXT or amblyopia (other than refractive correction) within the past 4 weeks, including vision therapy, orthoptics, patching, atropine, or other penalization
* Substantial overminus spectacles (spectacles overminused by more than 1.00 D SE than the most recent cycloplegic refraction and also results in minus SE power in the spectacles; underplussing is allowed) within the past 4 weeks
* Prior strabismus, intraocular, or refractive surgery (including BOTOX injection)
* Previous use of prism spectacles

Additional Eligibility Criteria for Randomization Based on Prism Adaptation Testing

* Exodeviation by PACT while wearing "trial" relieving prism for 30 minutes is smaller at distance or near than measured during initial testing (e.g. not fully adapting to prism at both distances)
* No new esotropia on cover test at near while wearing "trial" relieving prism for 30 minutes, compared with enrollment measurement taken without prism
* No esodeviation >6 Δ on PACT at near while wearing "trial" relieving prism for 30 minutes

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David G Morrison, MD, Study Chair — Vanderbilt University Medical Center; Allison I Summers, OD, MCR, Study Chair — Oregon Health and Science University
Locations (28):
- United States (28):
  - UAB Pediatric Eye Care; Birmingham Health Care, Birmingham, Alabama
  - Midwestern University Eye Institute, Glendale, Arizona
  - Arkansas Childrens, Little Rock, Arkansas
  - Southern California College of Optometry, Fullerton, California
  - Western University College of Optometry, Pomona, California
  - Nova Southeastern University College of Optometry, The Eye Institute, Fort Lauderdale, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Illinois College of Optometry, Chicago, Illinois
  - University of Chicago, Hyde Park, Illinois
  - Indiana School of Optometry, Bloomington, Indiana
  - Indiana University School of Optometry, Indianapolis, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - University of Kentucky Department of Neurology, Lexington, Kentucky
  - Wilmer Eye Institute, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Boston Children's Hospital Waltham, Boston, Massachusetts
  - Pediatric Ophthalmology, P.C., Grand Rapids, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Ohio State University College of Optometry, Columbus, Ohio
  - OHSU Casey Eye Institute, Portland, Oregon
  - Pediatric Ophthalmology of Erie, Erie, Pennsylvania
  - Salus University/Pennsylvania College of Optometry, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Children's Hospital - Dept. Of Ophthalmology, Houston, Texas
  - Houston Eye Associates, The Woodlands, Texas
  - Virginia Pediatric Eye Center, Norfolk, Virginia
  - Gundersen Health System, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH data sharing policy, a de-identified database is placed in the public domain on the Pediatric Eye Disease Investigator Group (PEDIG) public website after the completion of each protocol and publication of the primary manuscript.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available after publication.
Access Criteria: Users accessing the data must enter an email address.
URL: http://pedig.jaeb.org

REFERENCES:
- [Result] Summers AI, Morrison DG, Chandler DL, Henderson RJ, Chen AM, Leske DA, Walker KR, Li Z, Melia BM, Bitner DP, Kurup SP, Allen M, Phillips PH, Nash DL, Grigorian AP, Kraus CL, Miller AM, Titelbaum JR, Kraker RT, Holmes JM, Cotter SA; Pediatric Eye Disease Investigator Group. A Pilot Randomized Clinical Trial of Base-in Relieving Prism Spectacle Treatment of Intermittent Exotropia. Optom Vis Sci. 2023 Jul 1;100(7):432-443. doi: 10.1097/OPX.0000000000002039. Epub 2023 Jul 1. PMID 37399233
- [Result] Hatt SR, Leske DA, Holmes JM, Henderson RJ, Chandler DL, Morrison DG, Summers AI, Cotter SA. Testing depth of suppression in childhood intermittent exotropia. J AAPOS. 2022 Feb;26(1):36-38.e1. doi: 10.1016/j.jaapos.2021.08.303. Epub 2021 Nov 16. PMID 34793970
- See also: PEDIG Public Website — https://public.jaeb.org/pedig

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 09/01/2019 and 07/30/2020, 61 participants were enrolled into the study across 28 clinical sites. After prism-adaptation testing to confirm eligibility, 4 participants did not meet eligibility criteria and 57 participants were randomized to receive either 40% base-in prism spectacles (n=28) or non-prism spectacles (n=29).
Pre-assignment Details: After enrollment testing and prior to randomization, an in-office prism adaptation test was administered so that children with "full" prism adaptation (i.e., deviation magnitude increases by the amount of prism worn) would be excluded from the trial. Of 61 participants enrolled, 4 participants did not meet eligibility criteria after prism-adaptation testing and were dropped prior to randomization.
Period: Overall Study
Arm/Group | Prism Group | Non-Prism Group
Started | 28 | 29
Completed | 25 | 25
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prism Group | Non-Prism Group | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28 | 29 | 57
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.4 (2.4) | 6.8 (2.1) | 6.6 (2.2)
Age, Customized [Count of Participants; unit: Participants]
  3 to <5 years | 10 | 7 | 17
  5 to <7 years | 7 | 10 | 17
  7 to <9 years | 8 | 8 | 16
  >=9 years | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 11 | 13 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 3 | 3
  Black/African American | 6 | 2 | 8
  Hispanic | 4 | 7 | 11
  White | 16 | 17 | 33
  More than one race | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 28 | 29 | 57
Refractive Error Average of Eyes, Continuous [Mean (Standard Deviation); unit: Spherical Equivalent Diopters] — Average spherical equivalent in diopters (D) of the right and left eye after cycloplegic refraction within 7 months of enrollment.
  Spherical Equivalent Diopters | 0.3 (1.0) | 0.1 (1.4) | 0.2 (1.2)
Refractive Error Average of Eyes, Categorical [Count of Participants; unit: Participants] — Average spherical equivalent in diopters (D) of the right and left eye after cycloplegic refraction within 7 months of enrollment.
  Participants
    -6.00 to <-2.00 diopters | 1 | 3 | 4
    -2.00 to <-1.00 diopters | 2 | 0 | 2
    -1.00 to <-0.00 diopters | 4 | 4 | 8
    0.00 to <1.00 diopters | 12 | 16 | 28
    1.00 to <2.00 diopters | 9 | 6 | 15
Treatment for Intermittent Exotropia Prior to Enrollment [Count of Participants; unit: Participants]
  Overminus Lenses | 2 | 3 | 5
  Patching | 7 | 5 | 12
  Patching and Atropine | 0 | 1 | 1
  Patching and Overminus Lenses | 1 | 0 | 1
  Vision Therapy and Overminus Lenses | 0 | 1 | 1
  None | 18 | 19 | 37
Randot Preschool Stereoacuity at Near, Continuous [Mean (Standard Deviation); unit: log arcsec] — Randot® Preschool Stereoacuity test (Stereo Optical Co., Inc., Chicago, IL). For analysis, stereoacuity was converted from seconds of arc scores to log arcsec values (in parentheses) as follows: 40 (1.60), 60 (1.78), 100 (2.00), 200 (2.30), 400 (2.60), 800 (2.90); participants with no detectable (nil) stereoacuity were assigned the value of 1600 (3.20). A lower number is better.
  log arcsec | 2.3 (0.4) | 2.3 (0.5) | 2.3 (0.4)
Randot Preschool Stereoacuity at Near, Categorical [Count of Participants; unit: Participants] — Randot® Preschool Stereoacuity test (Stereo Optical Co., Inc., Chicago, IL). For analysis, stereoacuity was converted from seconds of arc scores to log arcsec values (in parentheses) as follows: 40 (1.60), 60 (1.78), 100 (2.00), 200 (2.30), 400 (2.60), 800 (2.90); participants with no detectable (nil) stereoacuity were assigned the value of 1600 (3.20). A lower number is better.
  Participants
    40 (1.60) | 2 | 3 | 5
    60 (1.78) | 6 | 8 | 14
    100 (2.00) | 9 | 7 | 16
    200 (2.30) | 3 | 4 | 7
    400 (2.60) | 5 | 3 | 8
    800 (2.90) | 2 | 2 | 4
    Nil (3.10) | 1 | 2 | 3
Suppression [Count of Participants; unit: Participants] — The suppression assessment is a standardized method of assessing the depth of suppression experienced while the participant is tropic (NOT aligned). Scoring is reported on an ordinal scale from 0 (no suppression) to 3 (dense suppression). "Missing" refers to cases in which participants were unable to understand the test and/or gave unreliable responses.
  Participants
    None (0 suppression) | 3 | 3 | 6
    Mild (1 suppression) | 1 | 4 | 5
    Moderate (2 suppression) | 4 | 8 | 12
    Dense (3 suppression) | 18 | 10 | 28
    Missing | 2 | 4 | 6
Exotropia Control Score at Distance, Continuous [Mean (Standard Deviation); unit: units on a scale] — Control of the exodeviation was measured at distance using the IXT Office Control Score, (Mohney, 2006) which ranges from 0 (phoria) to 5 (constant exotropia). Control levels 3-5 were assigned based on the duration of manifest exotropia during a 30-second period before any dissociation. If no exotropia was observed, control levels 0-2 were assigned based on the longest time to reestablishing fusion after 3 consecutive 10-second periods of dissociation. Control was measured at the beginning, middle, and end (3 tests) of a 20- to 40-minute office examination, and the mean was used.
  units on a scale | 3.4 (0.9) | 3.5 (0.9) | 3.5 (0.9)
Exotropia Control Score at Near, Continuous [Mean (Standard Deviation); unit: units on a scale] — Control of the exodeviation was measured at near using the IXT Office Control Score, (Mohney, 2006) which ranges from 0 (phoria) to 5 (constant exotropia). Control levels 3-5 were assigned based on the duration of manifest exotropia during a 30-second period before any dissociation. If no exotropia was observed, control levels 0-2 were assigned based on the longest time to reestablishing fusion after 3 consecutive 10-second periods of dissociation. Control was measured at the beginning, middle, and end (3 tests) of a 20- to 40-minute office examination, and the mean was used.
  units on a scale | 2.3 (1.3) | 1.7 (1.1) | 2.0 (1.2)
Exotropia Control Score at Distance, Categorical [Count of Participants; unit: Participants] — Mean of 3 assessments performed throughout exam. Mean distance exotropia control of 2 points or greater (worse) was required for eligibility.
  Participants
    0 to <1 unit | 0 | 0 | 0
    1 to <2 units | 0 | 0 | 0
    2 to <3 units | 8 | 8 | 16
    3 to <4 units | 10 | 10 | 20
    4 to 5 units | 10 | 11 | 21
Exotropia Control Score at Near, Categorical [Count of Participants; unit: Participants] — Mean of 3 assessments performed throughout exam. Mean near exotropia control of less than 5 points (i.e., could not be constant on all 3 measures) was required for eligibility.
  Participants
    0 to 1 unit | 2 | 6 | 8
    1 to <2 units | 9 | 9 | 18
    2 to <3 units | 6 | 9 | 15
    3 to <4 units | 6 | 4 | 10
    4 to 5 units | 5 | 1 | 6
Exodeviation by PACT at Distance, Categorical [Count of Participants; unit: Participants] — Eligibility criteria: Distance exodeviation at least 16∆ measured by PACT and no larger than 35∆. Near deviation does not exceed the distance deviation by more than 10∆ by PACT. A higher deviation is worse.
  Participants
    1 to 9 pd | 0 | 0 | 0
    10 to 15 pd | 0 | 0 | 0
    16 to 18 pd | 3 | 5 | 8
    20 to 25 pd | 18 | 15 | 33
    30 to 35 pd | 7 | 9 | 16
    40 to 45 pd | 0 | 0 | 0
Exodeviation by PACT at Distance, Continuous [Mean (Standard Deviation); unit: Prism Diopters (pd)] — Eligibility criteria: Distance exodeviation at least 16∆ measured by PACT and no larger than 35∆. Near deviation does not exceed the distance deviation by more than 10∆ by PACT. A higher deviation is worse.
  Prism Diopters (pd) | 25.1 (4.7) | 24.9 (5.6) | 25.0 (5.2)
Exodeviation by PACT at Near, Categorical [Count of Participants; unit: Participants] — Eligibility criteria: Near exodeviation at least 10∆ measured by PACT and no larger than 35∆. Near deviation does not exceed the distance deviation by more than 10∆ by PACT. A higher deviation is worse.
  Participants
    1 to 9 pd | 0 | 0 | 0
    10 to 15 pd | 2 | 6 | 8
    16 to 18 pd | 8 | 7 | 15
    20 to 25 pd | 15 | 8 | 23
    30 to 35 pd | 3 | 8 | 11
    40 to 45 pd | 0 | 0 | 0
Exodeviation by PACT at Near, Continuous [Mean (Standard Deviation); unit: Prism Diopters (pd)] — Eligibility criteria: Near exodeviation at least 10∆ measured by PACT and no larger than 35∆. Near deviation does not exceed the distance deviation by more than 10∆ by PACT. A higher deviation is worse.
  Prism Diopters (pd) | 21.5 (5.1) | 21.1 (7.5) | 21.3 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Exotropia Control Score at Distance, Continuous Score
Description: The primary analysis will be an intent-to-treat comparison of mean 8-week control of the distance exodeviation (average of 3 measurements) between treatment groups using an analysis of covariance (ANCOVA) model, which adjusts for baseline distance control. Distance control scores range from 0 to 5 with higher scores indicating a worse outcome.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 25 | 25
units on a scale | 3.6 (1.3) | 3.3 (1.5)
Statistical Analysis 1: Comparison: Prism Group vs Non-Prism Group; The primary analysis was the treatment group difference (and 95% CI) in mean distance control at the 8-week outcome visit using an ANCOVA adjusted for baseline distance control. The planned convenience sample size of 64 was expected to provide outcome data for at least 60 participants (30 per group); Test type: Superiority; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.5 to 1.1] — Difference in mean control and 95% confidence interval (CI) are from ANCOVA model adjusting for corresponding baseline control score. Prism group minus Non-Prism group (positive difference indicates Prism group worse than Non-Prism group)

2. Secondary Outcome: Exotropia Control Score at Distance, % With Treatment Response
Description: The secondary analysis will calculate the percentage of participants with a "treatment response," defined as ≥1 point improvement in control of their distance exodeviation (average of 3 measurements) between baseline and the 8-week outcome exam.
Time Frame: 8 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 25 | 25
percentage of participants | 32 | 24
Statistical Analysis 1: Comparison: Prism Group vs Non-Prism Group; Test type: Superiority; Mean Difference (Final Values) = 8, 95% CI 2-sided [-17 to 32] — Difference between Prism minus Non-Prism group (positive difference indicates Prism group better than Non-Prism group)

3. Secondary Outcome: Exotropia Control Score at Distance and Near, % With No Spontaneous Tropia
Description: The proportion of participants with no spontaneous tropia at 8 weeks will be compared between treatment groups using a two-sided Barnard's test with alpha of 0.05, with calculation of a two-sided 95% confidence interval on the difference in proportions.
  No spontaneous tropia at the 8-week primary outcome exam is defined as a score of ≤2 (0, 1, or 2) on all three assessments of control at distance and at near.
Time Frame: 8 Weeks
Measure: Number; unit: percentage of participants
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 25 | 25
percentage of participants | 48 | 51
Statistical Analysis 1: Comparison: Prism Group vs Non-Prism Group; Test type: Superiority; Mean Difference (Final Values) = -4, 95% CI 2-sided [-27 to 19] — Difference between Prism minus Non-Prism group (positive difference indicates Prism group better than Non-Prism group)

4. Secondary Outcome: Exotropia Control Score at Distance, Continuous Change Between Baseline and 8 Weeks
Description: Control of the exodeviation was measured at distance using the IXT Office Control Score, (Mohney, 2006) which ranges from 0 (phoria) to 5 (constant exotropia). Control levels 3-5 were assigned based on the duration of manifest exotropia during a 30-second period before any dissociation. If no exotropia was observed, control levels 0-2 were assigned based on the longest time to reestablishing fusion after 3 consecutive 10-second periods of dissociation. Control was measured at the beginning, middle, and end (3 tests) of a 20- to 40-minute office examination, and the mean was used. The change in distance control from baseline to 8 weeks will be calculated. A negative value indicates improvement.
Time Frame: 8 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 25 | 25
units on a scale | 0.1 (1.4) | -0.2 (1.5)

5. Secondary Outcome: Exotropia Control Score at Near, Continuous Score
Description: Near control will be evaluated similarly to the primary outcome and outcome measures 2-4. Near control scores range from 0 to 5 with higher scores indicating a worse outcome.
Time Frame: 8 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 25 | 25
units on a scale | 1.7 (1.1) | 1.7 (1.3)
Statistical Analysis 1: Comparison: Prism Group vs Non-Prism Group; The secondary analysis was the treatment group difference (and 95% CI) in mean near control at the 8-week outcome visit using an ANCOVA adjusted for baseline near control; Test type: Superiority; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.7 to 0.7] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Exodeviation by PACT at Distance, Continuous
Description: The measure of ocular alignment at distance by PACT will be summarized at 8 weeks for each treatment group. A higher deviation is worse.
Time Frame: 8 Weeks
Measure: Mean (Standard Deviation); unit: prism diopters
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 25 | 25
prism diopters | 30.6 (9.3) | 26.5 (8.1)

7. Secondary Outcome: Exodeviation by PACT at Near, Continuous
Description: The measure of ocular alignment at near by PACT will be summarized at 8 weeks for each treatment group. A higher deviation is worse.
Time Frame: 8 Weeks
Measure: Mean (Standard Deviation); unit: prism diopters
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 25 | 25
prism diopters | 28.7 (8.2) | 19.0 (9.8)

8. Secondary Outcome: Randot Preschool Stereoacuity at Near, Continuous
Description: Randot® Preschool Stereoacuity test (Stereo Optical Co., Inc., Chicago, IL). For analysis, stereoacuity was converted from seconds of arc scores to log arcsec values (in parentheses) as follows: 40 (1.60), 60 (1.78), 100 (2.00), 200 (2.30), 400 (2.60), 800 (2.90); participants with no detectable (nil) stereoacuity were assigned the value of 1600 (3.20). The measure of Randot Preschool Stereoacuity at near will be summarized at 8 weeks for each treatment group. A lower score is better.
Time Frame: 8 Weeks
Measure: Mean (Standard Deviation); unit: log arc seconds
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 25 | 25
log arc seconds | 2.2 (0.4) | 1.9 (0.4)

9. Secondary Outcome: Compliance of Spectacle Wear
Description: Parents will be asked to complete a compliance calendar by recording the percentage of time their child has worn the study-prescribed spectacle correction each day. Proportion of time worn each day will be described as excellent (76% to 100%), good (51% to 75%), fair (26% to 50%), poor (1 to 25%), or none (0%). Based on review of the calendars and discussion with parents at the 8-week outcome exam, the investigator will record the total proportion of time worn as excellent (76% to 100%), good (51% to 75%), fair (26% to 50%), poor (1 to 25%), or none (0%: did not fill prescription or never picked up spectacles).
  The distribution of compliance will be assessed for each treatment group at the outcome exam.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 25 | 25
Participants
  Excellent (76% to 100%) | 22 | 22
  Good (51% to 75%) | 3 | 2
  Fair (26% to 50%) | 0 | 1
  Poor (1% to 25%) | 0 | 0
  None (0%) | 0 | 0

10. Secondary Outcome: Child Assessment of Symptoms - Do Your Eyes Hurt?
Description: Adverse symptoms of intermittent exotropia will be summarized at the 8-week outcome exam using a symptom survey that is administered to the child. Response options are based on frequency of observations: never, sometimes, and always. The distribution of scores on each survey item will be tabulated by treatment group after 8-weeks.
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 25 | 25
Participants
  Never | 15 | 22
  Sometimes | 6 | 3
  Almost Always | 4 | 0

11. Secondary Outcome: Child Assessment of Symptoms - Do Your Eyes Feel Funny?
Description: as for outcome 10
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 25 | 25
Participants
  Never | 17 | 20
  Sometimes | 7 | 3
  Almost Always | 1 | 2

12. Secondary Outcome: Child Assessment of Symptoms - Do You Have Double Vision?
Description: as for outcome 10
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 25 | 25
Participants
  Never | 17 | 17
  Sometimes | 8 | 7
  Almost Always | 0 | 1

13. Secondary Outcome: Child Assessment of Symptoms - Is it Hard for You to Stare at Things?
Description: as for outcome 10
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 25 | 25
Participants
  Never | 16 | 15
  Sometimes | 7 | 8
  Almost Always | 2 | 2

14. Secondary Outcome: Child Assessment of Symptoms - Do You Have Problems With Your Eyes in the Sun?
Description: as for outcome 10
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 25 | 25
Participants
  Never | 11 | 14
  Sometimes | 8 | 5
  Almost Always | 6 | 6

15. Secondary Outcome: Child Assessment of Symptoms - Do Your Eyes go in and Out?
Description: as for outcome 10
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 25 | 25
Participants
  Never | 20 | 19
  Sometimes | 2 | 3
  Almost Always | 3 | 3

16. Secondary Outcome: Child Assessment of Symptoms - Is it Hard to Focus Your Eyes?
Description: as for outcome 10
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 25 | 25
Participants
  Never | 16 | 12
  Sometimes | 5 | 11
  Almost Always | 4 | 2

17. Secondary Outcome: Parent Assessment of Symptoms and Spectacle Wear - Has Your Child Had Headaches?
Description: Adverse symptoms of intermittent exotropia and spectacle wear will be summarized at the 8-week outcome exam using a symptom survey that is administered to the parent.
  Response options are based on frequency of observations: never, almost never, sometimes, often, and almost always. The distribution of scores on each survey item will be tabulated by treatment group after 8-weeks.
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 25 | 25
Participants
  Never | 15 | 14
  Almost Never | 8 | 6
  Sometimes | 2 | 5
  Often | 0 | 0
  Almost Always | 0 | 0

18. Secondary Outcome: Parent Assessment of Symptoms and Spectacle Wear - Has Your Child Had Eyestrain?
Description: as for outcome 17
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 25 | 25
Participants
  Never | 16 | 11
  Almost Never | 5 | 4
  Sometimes | 4 | 9
  Often | 0 | 1
  Almost Always | 0 | 0

19. Secondary Outcome: Parent Assessment of Symptoms and Spectacle Wear - Has Your Child Avoided Reading or Doing Things up Close?
Description: as for outcome 17
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 25 | 25
Participants
  Never | 22 | 15
  Almost Never | 2 | 6
  Sometimes | 0 | 3
  Often | 1 | 1
  Almost Always | 0 | 0

20. Secondary Outcome: Parent Assessment of Symptoms and Spectacle Wear - Has Your Child Reported Blurry Vision?
Description: as for outcome 17
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 25 | 25
Participants
  Never | 21 | 21
  Almost Never | 2 | 3
  Sometimes | 1 | 1
  Often | 1 | 0
  Almost Always | 0 | 0

21. Secondary Outcome: Parent Assessment of Symptoms and Spectacle Wear - Has Your Child Looked Over His or Her Spectacles?
Description: as for outcome 17
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 25 | 25
Participants
  Never | 12 | 14
  Almost Never | 7 | 3
  Sometimes | 5 | 5
  Often | 0 | 3
  Almost Always | 1 | 0

22. Secondary Outcome: Parent Assessment of Symptoms and Spectacle Wear - Has Your Child Taken His/Her Spectacles Off When he/She Should be Wearing Them?
Description: as for outcome 17
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 25 | 25
Participants
  Never | 5 | 10
  Almost Never | 11 | 5
  Sometimes | 6 | 8
  Often | 3 | 1
  Almost Always | 0 | 1

23. Secondary Outcome: Parent Assessment of Symptoms and Spectacle Wear - Has Your Child Complained That the Spectacles Hurt His/Her Ears and/or Nose?
Description: as for outcome 17
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 25 | 25
Participants
  Never | 17 | 14
  Almost Never | 3 | 5
  Sometimes | 5 | 5
  Often | 0 | 1
  Almost Always | 0 | 0

24. Other Pre Specified Outcome: Distance Visual Acuity (Snellen Equivalent)
Description: Distance visual acuity will be assessed at the 8-week outcome exam. Any optotype method can be used for testing. The distribution of distance visual acuity Snellen Equivalents will be tabulated for each treatment group. A lower Snellen Equivalent is best.
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 25 | 25
Participants
  20/16 (best) | 3 | 1
  20/20 | 10 | 9
  20/25 | 9 | 8
  20/32 | 2 | 3
  20/40 | 1 | 4

25. Other Pre Specified Outcome: Fusional Convergence - Continuous Break Point
Description: As an exploratory analysis, the distribution of fusional convergence amplitude (break point, blur point, and recovery) at 8 weeks will be summarized for each treatment group. Fusional amplitudes are a measure of how well a participant can converge their eyes using fusional vergence. It is measured by increasing base-out prism to the point that the participant is no longer able to control the deviation. The total amount of fusion is the magnitude of the base-out prism the participant was able to overcome plus the magnitude of the deviation. A higher number of prism diopters for break point is better than a lower number. A lower number for recovery point is better than a higher number.
Time Frame: 8 Weeks
Population: 3 participants in the Prism group and 2 participants in the Non-Prism group were unable to perform testing at 8 weeks and are not included.
Measure: Mean (Standard Deviation); unit: prism diopters
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 22 | 23
prism diopters | 17.8 (11.5) | 17.5 (10.9)

26. Other Pre Specified Outcome: Suppression
Description: The suppression assessment is a standardized method of assessing the depth of suppression experienced while the participant is tropic (NOT aligned). Scoring is reported on an ordinal scale from 0 (no suppression) to 3 (dense suppression). "Missing" refers to cases in which participants were unable to understand the test and/or gave unreliable responses. As an exploratory analysis, the distribution of suppression level (none, mild, moderate, severe, missing) will be tabulated after 8 weeks by treatment group.
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 25 | 25
Participants
  None (0 suppression) | 1 | 5
  Mild (1 suppression) | 5 | 3
  Moderate (2 suppression) | 6 | 4
  Dense (3 suppression) | 12 | 10
  Missing | 1 | 3

27. Other Pre Specified Outcome: Fusional Convergence - Continuous Recovery Point
Description: As an exploratory analysis, the distribution of fusional convergence amplitude (break point, blur point, and recovery) at 8 weeks will be summarized for each treatment group. Fusional amplitudes are a measure of how well a participant can converge their eyes using fusional vergence. It is measured by increasing base-out prism to the point that the participant is no longer able to control the deviation. The total amount of fusion is the magnitude of the base-out prism the participant was able to overcome plus the magnitude of the deviation. A higher number of prism diopters for break point is better than a lower number. A lower number for recovery is better than a higher number.
Time Frame: 8 Weeks
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: prism diopters
Arm/Group | Prism Group | Non-Prism Group
Number analyzed (Participants) | 22 | 23
prism diopters | 9.4 (10.1) | 10.6 (9.4)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/assessed from the participant's perspective between randomization and completion of their 8-week primary outcome visit.
Description: No adverse events are anticipated as a result of prism therapy or non-prism spectacle wear. No surgical procedures are part of the protocol and no treatments are being prescribed that are not part of usual care. Symptom survey data have been reported as outcomes by treatment group.
Arm/Group | Prism Group | Non-Prism Group
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29
Other Adverse Events (participants affected / at risk) | 0/28 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/70/NCT03998670/Prot_001.pdf
  • Statistical Analysis Plan (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/70/NCT03998670/SAP_002.pdf
  • Informed Consent Form (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT03998670/ICF_000.pdf